CLINICAL TRIAL: NCT05404763
Title: Evolution of Physical Activity in Severe Asthmatic Patients Treated With Mepolizumab
Brief Title: Mepolizumab and Physical Activity in Severe Asthma
Acronym: TEXAS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020_56; 2021-A03205-36 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-03-21; First posted 2022-06-03 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Asthma; Asthma; Eosinophilic
Keywords: Severe asthma,; Physical activity; Exercise; Dyspnea
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia; Motor Activity; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Severe asthma is a debilitating condition associated with frequent symptoms, life-threatening exacerbations and corticosteroid side-effects. Exercise limitation due to exercise-induced bronchoconstriction, dynamic lung hyperinflation and comorbidity may be a strong determinant of the disease burden. Mepolizumab is a monoclonal anti-interleukin-5 (IL-5) antibody that reduces the rate of severe exacerbations, asthma symptoms and oral glucocorticoid requirement, and improves quality of life and work productivity in severe eosinophilic asthma. However, its impact on physical activity and exercise tolerance is unknown. We hypothesize that a 6-month treatment with mepolizumab is associated with an improvement in daily life physical activity and exercise tolerance in relation with enhanced ventilatory mechanics.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years at the time of inclusion
* Asthma diagnosed for at least one year including a history of

  1. FEV1 and/or FVC reversibility of more than 12% and than 200 ml documented in the patient's record
  2. OR FEV1 variability of more than 20% between two visits
  3. OR positive methacholine test
* Severe uncontrolled asthma monitored for at least six months in the investigation center with at least two assessments:

  1. high-dose of inhaled corticosteroids (ICS >1,000 μg/day of beclometasone equivalent) in combination with another controller at a stable dosage for at least three months
  2. ACQ-5 score >1.5 and/or more than two severe exacerbations (i.e exacerbation requiring ≥ 3 days of systemic corticosteroids, hospitalization or admission at the emergency department) in the past year
  3. Blood eosinohils ≥300/mm3 within the 12 past months
  4. Decision to introduce mepolizumab according to regulatory approval
  5. Patient agreement to receive Mepolizumab
* Body mass index (BMI) within the range [18.5 - 35] kg/m2.
* Able to give signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol

Exclusion Criteria:

* Body Mass Index <18.5 or >35 kg/m2
* Active smoker or active smoking during the last 6 months or cumulative > 10 pack-years
* All conditions responsible for physical disability (neurological, orthopedic, psychiatric, non-exhaustive list) or other condition limiting exercise in the investigator's opinion
* Any chronic respiratory or cardiac pathology which may interfere with the assessment of asthma according to the investigator's opinion
* Prior treatment with mepolizumab or benralizumab
* Bronchial thermoplasty during the past 12 months
* Contraindication to mepolizumab
* Non-coverage by the social security insurance
* Pregnant, breastfeeding, or lactating women
* Patient unable to receive information
* Refusal to sign the consent form
* Unwillingness or inability to follow the study procedures, in the opinion of the investigator
* Person deprived of the liberty Person benefiting from a system of legal protection (guardianship…)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: uncontrolled eosinophilic severe asthma with indication for treatment with mepolizumab
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2025-02-02 (Estimated); Study Completion 2025-07-02 (Estimated)

PRIMARY OUTCOMES:
Number of daily steps | after 6 months of treatment with mepolizumab

SECONDARY OUTCOMES:
Time with moderate physical activity (between 3 and 6 METs) and intense activity (>6 METs) | Baseline, at 3 months and at 6 months
Percentage of time spent with moderate physical activity (between 3 and 6 METs) and intense activity (>6 METs) | Baseline, at 3 months and at 6 months
Ricci and Gagnon questionnaire score • | Baseline, at 3 months and at 6 months
  Ricci and Gagnon questionnaire is Score of physical activity , 9 items, total range score from 6 to 45, higher score indicating a higher level of physical activity
Endurance time during a sub-maximal exercise (80% of maximum load) | Baseline, at 3 months and at 6 months
Baseline Dyspnea Index (BDI) | Baseline, at 3 months and at 6 months
  The BDI is an interviewer-administered rating of severity of dyspnea at a single state. It provides a multidimensional measurement of dyspnea based on 3 components It comprises 3 domains (functional impairement, magnitude of task and magnitude of effort) scoring from 0 (very severe) to 4 (no impairment) with a recall of the last two weeks. The total score ranges from 0 to 12, the lower the score, the worse the severity of dyspnea.
Transition Dyspnea Index (TDI) scores | Baseline, at 3 months and at 6 months
  The TDI measures changes in each domain of dyspnea severity from the baseline as established by the BDI. The change is rated by seven grades ranging from -3 (major deterioration) to +3 (major improvement). The total score ranges from - 9 to + 9
The modified Medical Research Council (mMRC) scale | Baseline, at 3 months and at 6 months
  The mMRC scale is a self-assessed unidimensional scale rating the impact of dyspnea on physical activity in everyday life. The patient chooses the answer that best describes his level of limitation related to dyspnea among 5 proposals. The score is between 0 (absence of dyspnea) to 4 (permanent dyspnea). The MCID considered is 1 unit although data are limited.
Multidimensional Dyspnea Profile (MDP) scores | Baseline, at 3 months and at 6 months
  The MDP questionnaire is an 11-item hetero-questionnaire evaluating both sensory and affective dimensions of dyspnea, respectively the sensation produced by the respiratory stimulus and the emotion associated with this sensation.
ACQ-5 score | Baseline, at 3 months and at 6 months
  The ACQ-5 is a shortened version of the ACQ that assesses asthma symptoms (night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing) omitting the forced expiratory volume in 1 second measurement and short acting beta antagonist use from the original ACQ score. Patients are asked to recall how their asthma has been during the previous week by responding to 5 symptom questions. Questions are weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ-5 score is the mean of the responses. Mean scores of ≤0.75 indicate well-controlled asthma, scores between 0.75 and <1.5 indicate partly controlled asthma, and a score ≥1.5 indicates not well controlled asthma . Individual changes of at least 0.5 are considered to be clinically meaningful.
AQLQ score | Baseline, at 3 months and at 6 months
  The Asthma Quality of Life Questionnaire (AQLQ) is a 32-item, 4-domain instrument that can either be self- or interviewer-administered. The recall-time is two weeks. The four domains covered are: (i) symptoms (11 items), (ii) activity limitation (12 items, 5 of which are individualized), (iii) emotional function (5 items), and (iv) environmental exposure (4 items). Each item is ranked by the patient using a 7-point Likert scale ranging from 1 (severely impaired) to 7 (not impaired at all). Scores range from 1 to 7, higher scores indicate better quality of life and a minimally important difference (for overall scores and for each sub-domain) has been established at 0.5.
Hospital Anxiety and Depression scores (HADS) | Baseline, at 3 months and at 6 months
  Depressive symptoms will be assessed using The Hospital Depression and Anxiety Scale.The scale allows to detect anxiety and depression using 14 items rated from 0-3.
Respiratory capacity by Spirometry | Baseline, at 3 months and at 6 months
Respiratory capacity by plethysmography | Baseline, at 3 months and at 6 months
Forced inspiratory by Spirometry | Baseline, at 3 months and at 6 months
Ventilatory function by Spirometry | Baseline, at 3 months and at 6 months
Forced oscillation by impulse oscillometry (the Tremoflo ® oscillometry system) | Baseline, at 3 months and at 6 months
Frequency of serious and non-serious side effects | Baseline, at 3 months and at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Chenivesse, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Lille University Hospital, Lille, France